CLINICAL TRIAL: NCT04553263
Title: Relapse Prevention in Stimulant Use Disorder
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study never initiated
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Edythe London, Professor of Psychiatry and Biobehavioral Sciences and Molecular and Medical Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-001075
Record Dates: First submitted 2020-06-03; First posted 2020-09-17 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Stimulant Use; Relapse; Cognitive Function; ADHD
Keywords: Stimulant Abuse; Relapse Prevention; ADHD; Contrave; Bupropion
MeSH Terms: conditions — Recurrence; Attention Deficit Disorder with Hyperactivity | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Contrave (Experimental): Participants will receive daily weight loss medication, Contrave, at a dose of 360 mg (Naltrexone HCl 32mg, Bupropion HCl 360mg). The dose will be titrated: 8 mg/90 mg on Week 1, 16 mg/180 mg on Week 2, 24 mg/270 mg on Week 3 and 32 mg/360 mg on Week 4. Dosing will continue for a total of 4 weeks during inpatient treatment, and thereafter for another month, with compliance monitored by smartphone.
  Interventions: Drug: Contrave 8Mg-90Mg Extended-Release Tablet
- Bupropion (Experimental): Participants will receive daily extended-release oral bupropion (Wellbutrin XL) at a dose of 450 mg. The dose will be titrated: 150 mg on Days 1 and 2, 300 mg on Days 3 and 4, and 450 mg on Day 5. Dosing will continue for a total of 4 weeks during inpatient treatment, and thereafter for another month, with compliance monitored by smartphone. A reduction to 300 mg will permitted to alleviate medication-related adverse effects if they occur.
  Interventions: Drug: Bupropion
- Treatment As Usual (No Intervention): Participants will complete inpatient treatment as usual and will not receive any medication. This arm serves as a TAU control to compare outcomes versus Bupropion and Contrave arms.

INTERVENTIONS:
Drug: Contrave 8Mg-90Mg Extended-Release Tablet — Naltrexone HCl/Bupropion HCl is an FDA-approved weight-loss medication with efficacy via the mesolimbic dopamine system to reduce hunger and help control cravings.
  Other Names: Naltrexone HCl/Bupropion HCl 8 Mg-90 Mg
  Arms: Contrave
Drug: Bupropion — Bupropion is FDA-approved and marketed both as an antidepressant agent (Wellbutrin®) and treatment for smoking cessation (Zyban®) and has shown efficacy in reducing symptoms of depression and drug craving in stimulant users. it is also a promising candidate to improve cognition function.
  Other Names: Wellbutrin; Zyban
  Arms: Bupropion

SUMMARY:
The purpose of this study is to assess the relationship between bupropion, stimulant use and relapse, ADHD (Attention Deficit Hyperactivity Disorder), and measures of mood, drug craving, and inhibitory control in individuals enrolled in inpatient treatment for stimulant-use disorder with and without ADHD.

The experimenters hypothesize that Bupropion and Contrave (Bupropion/Naltrexone) will increase inhibitory control and decrease drug craving and depressive symptoms in recently abstinent stimulant users in inpatient treatment with effects greater than those seen in recently abstinent stimulant users completing inpatient treatment as usual. An additional hypothesis is that relapse rates after leaving inpatient treatment in the group receiving bupropion will be lower than those of the group completing inpatient treatment as usual.

The study design consists of four assessments of drug craving, inhibitory control, impulsive choice, and mood (depression and anxiety). The timepoints for these assessments include: A. baseline after entering treatment B. 2 weeks after starting drug C. 8 weeks after starting drug, and D. 1 month after leaving treatment. Following eligibility screening, 60 stimulant users will be enrolled in one of 3 groups. Group 1 Bupropion Active Group: 20 subjects will receive bupropion for 8 weeks during inpatient treatment. Group 2 Contrave Active Group: 20 subjects will receive Contrave for 8 weeks during inpatient treatment. Group 3 Control Group: 20 subjects enrolled in inpatient treatment will complete treatment as usual as well as the four assessments (A-D) described above but will not receive drug (convenience control). Half of the subjects in each group will be diagnosed with ADHD and half will not, for a total of 10 subjects per group with ADHD.

DETAILED DESCRIPTION:
1. Participants will be recruited from the Clare Foundation (CLARE|MATRIX), where they will be residing in a residential substance use disorder program. Potential participants recently admitted with stimulant use disorder will be given a flyer/research information sheet describing the study when they are admitted to the study. Interested parties will sign their name on the sheet to indicate their interest, and will meet with a UCLA research associate at Clare to discuss details of the protocol and undergo initial screening following verbal consent. Initial screening involves a one page screening sheet and discussing the information sheet with the research associate at Clare.
2. If participants remain eligible following initial screening, they will enroll in the study and the UCLA research associate will set up an in person screening to sign the informed consent form and undergo additional screening. After completing informed consent and going through the informed consent quiz, a Nurse Practitioner or physician will take a medical history, take a personal and family health profile, perform a physical examination (History & Physical). Participants who provide written consent will complete questionnaires about their mood, medical, psychiatric and drug use history, personality and life experiences. The screening visit will also include a psychiatric diagnostic interview (MINI International Neuropsychiatric Interview M.I.N.I) completed by a trained diagnostician. Participants will also give a urine sample to determine what drugs they have recently used, a breath sample to determine the carbon monoxide levels in their system. Participants will travel to UCLA to give a blood sample to assess complete blood count, metabolic panel, screening for infectious diseases (Hepatitis B and C, HIV, syphilis) and tests of kidney function and receive an ECG (electrocardiogram). After all screening procedures have been completed, a study physician will collect and review ECG and laboratory tests to determine eligibility.
3. After completing all screening procedures, eligible participants will complete the following baseline assessments:

   A) Visit 1:

   i. Prior to completing cognitive tasks behavioral testing, participants will will have their blood drawn by a London laboratory phlebotomist or will visit the Clinical and Translational Research Center (CTRC), where a registered nurse will draw approximately 40mL of blood. Blood samples will be assayed for genetic markers associated with smoking and stimulant use. The purpose of the genetic analysis is to examine the relationship between genetic polymorphisms, treatment outcomes, circulating study drug, and measures of cognitive function.

   The DNA (deoxyribonucleic acid) samples acquired from this protocol will be added to a larger database of DNA samples collected from participants in London Laboratory protocols. DNA samples will be stored for future use other than the aims and goals of this study. Participants will not receive their results because our laboratory is only qualified for genetic analyses associated with research purposes and is not certified for clinical assessment of genetic information.

   This blood sample will also be used to determine follicular and luteal phase in female participants.

   ii. Urine toxicology: Participants will provide urine to assess recent use of drugs.

   iii. Cognitive/behavioral testing: Participants will complete some of the following tasks to assess inhibitory control and decision-making: Working memory (N-back test), declarative memory (Rey Auditory Verbal Learning Task), sustained attention (Rapid Visual Information Processing), inhibitory control (Stop Signal Test) reward-based decision-making (Monetary Delay Discounting and Reversal Learning, BART [Balloon Analogue Risk Task], ART [Angling Risk Task]), and impulsive and risk taking behavior (BIS [Barratt Impulsiveness Scale], Willingness-to-wait task, Domain-Specific Risk-Taking (DOSPERT) Scale, UPPS-P Impulsive Behavior Scale, TCI [Temperament Character Inventory]), Loss Aversion, the Risk and Ambiguity Task, craving (Brief Meth Craving Questionnaire), mindfulness (Multidimensional Assessment of Interoceptive Awareness [MAIA], Mindful Attention Awareness Scale [MAAS], Body Perception Questionnaire Body Awareness Very Short Form [BPQ]), and withdrawal from cigarettes (Shiffman-Jarvik Withdrawal Scale) and amphetamines (Amphetamine Cessation Symptom Assessment [ASCA]).
4. Participants in the active medication pool will be assigned to Contrave or Bupropion treatment based on timing of entry into the study (the London laboratory will initially assess Contrave effects). Participants assigned to the convenience control group will complete treatment as usual and will not take medication. The medication conditions will require that participants take capsules as instructed over the course of 8 weeks. Medications for the upcoming week will be dispensed at the beginning of each week. At the end of each week, the participants will meet with the study physician for a check-up to monitor potential adverse events. After the 8-wk regimen, participants will undergo repeat testing cognitive and behavioral tests as described in section 3.

   Study Intervention and Procedures:

   All participants will receive inpatient treatment as usual, including cognitive behavioral therapy. Within 10 days of entering treatment, participants in Group 1 (Bupropion Group) will begin receiving daily extended-release oral bupropion (Wellbutrin XL) at a dose of 450 mg, which was well tolerated by individuals with methamphetamine use disorder in a prior study. The dose will be titrated: 150 mg on Days 1 and 2, 300 mg on Days 3 and 4, and 450 mg on Day 5. Dosing will continue for a total of 4 weeks during inpatient treatment, and thereafter for another month, with compliance monitored by smartphone. A reduction to 300 mg will permitted to alleviate medication-related adverse effects if they occur. Participants in Group 2 (Contrave Group) will begin receiving daily oral Contrave at a dose of 360 mg (Naltrexone HCl 32mg, Bupropion HCl 360mg), which was well tolerated by individuals in a prior study The dose will be titrated: 8 mg/90 mg on Week 1, 16 mg/180 mg on Week 2, 24 mg/270 mg on Week 3 and 32 mg/360 mg on Week 4. Dosing will continue for a total of 4 weeks during inpatient treatment, and thereafter for another month, with compliance monitored by smartphone.
5. After completing medication treatment (active) or treatment as usual (control), participants will complete the following assessments:

   A) Blood draw at UCLA in the final week of drug treatment - a blood sample will be taken to assess plasma levels of drug.

   B) Visit 2:

   i. Prior to completing cognitive tasks behavioral testing, participants will will have their blood drawn by a London laboratory phlebotomist or will visit the Clinical and Translational Research Center (CTRC), where a registered nurse will draw approximately 40mL of blood. Blood samples will be assayed for genetic markers associated with smoking and stimulant use. The purpose of the genetic analysis is to examine the relationship between genetic polymorphisms, treatment outcomes, circulating study drug, and measures of cognitive function.

   The DNA samples acquired from this protocol will be added to a larger database of DNA samples collected from participants in London Laboratory protocols. DNA samples will be stored for future use other than the aims and goals of this study. Participants will not receive their results because our laboratory is only qualified for genetic analyses associated with research purposes and is not certified for clinical assessment of genetic information.

   This blood sample will also be used to determine follicular and luteal phase in female participants.

   ii. Urine toxicology: Participants will provide urine to assess recent use of drugs.

   iii. Cognitive/behavioral testing: Participants will complete some of the following tasks to assess inhibitory control and decision-making: Working memory (N-back test), declarative memory (Rey Auditory Verbal Learning Task), sustained attention (Rapid Visual Information Processing), inhibitory control (Stop Signal Test) reward-based decision-making (Monetary Delay Discounting and Reversal Learning, BART, ART), and impulsive and risk taking behavior (BIS, Willingness-to-wait task, Domain-Specific Risk-Taking (DOSPERT) Scale, UPPS-P Impulsive Behavior Scale, TCI), Loss Aversion, the Risk and Ambiguity Task, craving (Brief Meth Craving Questionnaire), mindfulness (Multidimensional Assessment of Interoceptive Awareness [MAIA], Mindful Attention Awareness Scale [MAAS], Body Perception Questionnaire Body Awareness Very Short Form [BPQ]), and withdrawal from cigarettes (Shiffman-Jarvik Withdrawal Scale) and amphetamines (Amphetamine Cessation Symptom Assessment [ASCA]).
6. Follow-up visit - 1 month after exiting inpatient treatment, participants will return to UCLA to complete follow-up procedures assessing cognitive function and stimulant use.

A) Visit 3:

i. Prior to completing cognitive tasks behavioral testing, participants will will have their blood drawn by a London laboratory phlebotomist or will visit the Clinical and Translational Research Center (CTRC), where a registered nurse will draw approximately 40mL of blood. Blood samples will be assayed for genetic markers associated with smoking and stimulant use. The purpose of the genetic analysis is to examine the relationship between genetic polymorphisms, treatment outcomes, circulating study drug, and measures of cognitive function.

The DNA samples acquired from this protocol will be added to a larger database of DNA samples collected from participants in London Laboratory protocols. DNA samples will be stored for future use other than the aims and goals of this study. Participants will not receive their results because our laboratory is only qualified for genetic analyses associated with research purposes and is not certified for clinical assessment of genetic information.

This blood sample will also be used to determine follicular and luteal phase in female participants.

ii. Urine toxicology: Participants will provide urine to assess recent use of drugs.

iii. Cognitive/behavioral testing: Participants will complete some of the following tasks to assess inhibitory control and decision-making: Working memory (N-back test), declarative memory (Rey Auditory Verbal Learning Task), sustained attention (Rapid Visual Information Processing), inhibitory control (Stop Signal Test) reward-based decision-making (Monetary Delay Discounting and Reversal Learning, BART, ART), and impulsive and risk taking behavior (BIS, Willingness-to-wait task, Domain-Specific Risk-Taking (DOSPERT) Scale, UPPS-P Impulsive Behavior Scale, TCI), Loss Aversion, the Risk and Ambiguity Task, craving (Brief Meth Craving Questionnaire), mindfulness (Multidimensional Assessment of Interoceptive Awareness [MAIA], Mindful Attention Awareness Scale [MAAS], Body Perception Questionnaire Body Awareness Very Short Form [BPQ]), and withdrawal from cigarettes (Shiffman-Jarvik Withdrawal Scale) and amphetamines (Amphetamine Cessation Symptom Assessment [ASCA]).

iv. Stimulant use measurements: Participants will complete timeline followback and self-report assessments of their recent stimulant use.

ELIGIBILITY:
Inclusion Criteria:

1. English fluency (in order to provide informed consent and complete questionnaires)
2. Age of 18-65 years inclusive
3. Meeting DSM 5 criteria for Stimulant-use disorder
4. Being 2-8 weeks abstinent from drugs of abuse other than nicotine (in cigarettes)
5. Vital signs as follows: resting pulse between 50 and 95 bpm, blood pressures between 90-150 mm Hg systolic and 45-95 mm Hg diastolic (inclusive)
6. Hematology and chemistry laboratory test results within normal (+/- 20%) limits and/or indicative of normal kidney function (estimated glomerular filtration rate ≥ 90 ml/min/1.73 m2) and/or not indicative of active disorder or infection.
7. Baseline ECG demonstrating normal conduction (including QTc) without clinically significant arrhythmias
8. Absence of clinically significant contraindications for participation, in the judgment of the admitting physician and the principal investigator, assessed by a medical history and physical examination.
9. Entering into and remaining in treatment voluntarily.

Exclusion Criteria:

1. Age of <18 or >65 years.
2. Current or past history of seizure disorder, including alcohol- or stimulant-related seizure, or significant family history of idiopathic seizure disorder or conditions that increase seizure risk (arteriovenous malformation, severe head injury, CNS tumor, CNS infection, stroke, anorexia nervosa or bulimia (current or prior diagnosis), and current use of drugs that lower seizure threshold
3. Current severe substance use disorder assessed by the MINI on any psychoactive substance (e.g., opioids) other than methamphetamine, cocaine or nicotine, or have physiological dependence on alcohol or a sedative-hypnotic (e.g., a benzodiazepine) requiring medical detoxification, or undergoing abrupt discontinuation of ethanol or sedatives including anticonvulsants, barbiturates, or benzodiazepines
4. Prior therapy with any opiate-substitutes (methadone, LAAM, buprenorphine) within 2 months of enrollment.
5. Previous adverse reaction to Bupropion or Naltrexone.
6. Current use of a. Bupropion, Naltrexone, opiates or opiate-substitutes, stimulants b.Any medications that directly affect dopaminergic or serotonergic neurotransmission in brain (i.e., SNRI, MAO-I, TCA) c. Any neuroleptic agent d. Systemic corticosteroids, Xanthines (i.e., theophylline) e. Sympathomimetics f. Antiretrovirals (i.e., nelfinavir, ritonavir and efavirenz) g. Linezolid or IV methylene blue h. Warfarin
7. MAO-I use in the 2 weeks before enrollment
8. Disease or injury preventing use of both eyes and ability to complete computer tasks assessing cognitive function (e.g. glaucoma, colorblindness)
9. Brain injury with loss of consciousness >30 min
10. Pre-existing psychotic disorders, bipolar disorder, organic brain disorder, or dementia as assessed by the MINI interview, or medical disorder, any of which require an excluded medication (e.g., antidepressant, neuroleptic, systemic corticosteroid, xanthine) or which would make medication compliance difficult.
11. Electroconvulsive therapy within the 90 days before screening.
12. Current suicidal ideation or plan, as assessed by the MINI
13. Untreated or unstable medical illness including, but not limited to endocrine, autoimmune, renal, hepatic, active infectious disease (like active tuberculosis and active syphilis), diabetes or use of insulin, neurological disorders (including, but not limited to Parkinson's disease, dementia.), uncontrolled hypertension (See NIDA Guidelines on Hypertension in the Operations Manual), significant heart disease (including but not limited to angina, any ECG/cardiovascular abnormality e.g., QTc interval prolongation > 450 milliseconds in men or 480 milliseconds in women or myocardial infarction within one year of enrollment).
14. Pregnancy or lactation [Note: Female participants must be either postmenopausal or using a reliable form of contraception (e.g., abstinence, oral contraceptive pills, intrauterine device, sterilization, condoms or spermicide). Women must have negative urine tests for pregnancy at study entry and at every weekly session]
15. Diagnosis of adult (i.e., 21 years or older) asthma, or chronic obstructive pulmonary disease (COPD), including those with a history of acute asthma within the 2 years before enrollment, and current or recent (past 3 months) treatment with theophylline, or have an FEV1 <70 %.
16. Currently receiving HIV treatment with antiviral and/or non-antiviral therapy since these drugs may increase the bupropion levels. The following list of HIV treatment/medications may be used: Norvir, Reyataz, Truvada, Videx, Viread, Androgel and Trizovir. Note: Any HIV medication not on this list should be approved by the medical monitor.
17. Neurological disorder that would compromise informed consent or complicate data interpretation (e.g., organic brain disease or dementia).
18. Any condition that, as deemed by the investigators and study physician, would compromise safe participation.
19. Meeting the definition of "prisoner" status, as defined by 45 CFR 46.303(c). This will be determined by UCLA research associates in collaboration with counselors at the Clare Matrix to confirm legal issues. Initial eligibility will be determined upon entry into the treatment center based on information given by the subject when entering treatment and the criteria added to the screening sheet.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-11 (Estimated); Primary Completion 2025-01-11 (Estimated); Study Completion 2025-01-11 (Estimated)

PRIMARY OUTCOMES:
Stimulant use 1 month after leaving inpatient treatment (self-report) | 84 days
  Stimulant use 1 month after leaving inpatient treatment, assessed via self-report. toxicology
Stimulant use 1 month after leaving inpatient treatment (urine toxicology) | 84 days
  Stimulant use 1 month after leaving inpatient treatment, assessed via urine sample.

SECONDARY OUTCOMES:
Sustained attention | 84 days
  The Continuous Performance Task will be used to assess sustained attention at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment.
Working memory | 84 days
  The Sternberg Spatial task will be used to assess working memory at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment.
Declarative memory | 84 days
  The Rey Auditory Verbal Learning Test will be used to assess declarative memory at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment.
Inhibitory control - stop signal task | 84 days
  The Stop-signal task will be used to assess inhibitory control at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment.
Inhibitory control - reversal learning | 84 days
  A reversal learning task will be used to assess inhibitory control at at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment.
Reward-based decision-making | 84 days
  A monetary delay-discounting task and the Balloon Analogue Risk task will be used to assess reward-based decision-making at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment.
Decision making under risk and ambiguity | 84 days
  A task involving decision making under during differing types of risk and ambiguity will be used to determine decision making under risk and ambiguity at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment. This task does not have a more specific name but involves a computer program testing decision making while participants are aware and unaware of probabilities for the outcomes of their responses.
Loss Aversion | 84 days
  A computer task assessing loss preferences will be used to assess loss aversion at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment.

OTHER OUTCOMES:
Personality - impulsivity | 84 days
  Self-report of impulsivity will be measured at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment using the Barratt Impulsiveness Scale.
Personality - novelty seeking | 84 days
  Self-report of novelty seeking will be measured at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment using the Temperament and Character Inventory.
Personality - reward dependence | 84 days
  Self-report of reward dependence will be measured at baseline prior to Contrave/Bupropion/placebo, after 8 weeks of Contrave/Bupropion/placebo treatment and 1 month after leaving inpatient treatment using the Temperament and Character Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Edythe D London, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States